CLINICAL TRIAL: NCT02173145
Title: Azithromycin for the Treatment of Cough in Idiopathic Pulmonary Fibrosis- a Clinical Trial
Brief Title: Azithromycin in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 002/14
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Idiopathic Pulmonary Fibrosis; Cough
Keywords: idiopathic pulmonary fibrosis; cough; immunomodulation; macrolide
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cough | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin first, Placebo second (Active Comparator): Medication with Azithromycin 500mg/d 3x/week p.o. o.d. for 12 weeks or placebo.
  Interventions: Drug: azithromycin; Drug: placebo
- Placebo first, Azithromycin second (Active Comparator): Medication with Azithromycin 500mg/d 3x/week p.o. o.d. for 12 weeks or placebo. Placebo will be capsulated similar to verum and given 3 times a week.
  Interventions: Drug: azithromycin; Drug: placebo

INTERVENTIONS:
Drug: azithromycin — Azithromycin is a macrolide antibiotic. 500mg Azithromycin will be given p.o. 3 times a week for 3 months. Azithromycin will be compared to placebo.
Drug: placebo — Placebo will be given 3 times a wek over a period of 3 months.

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a devastating disease with no cure available. Patients suffer from respiratory symptoms including dyspnea and cough. To improve life quality the investigators will test the effects of immunomodulation of macrolides specifically on cough in IPF patients. The investigators hypothesize that immunomodulatory treatment reduces cough frequency and might improve lung function.

DETAILED DESCRIPTION:
Background

Idiopathic pulmonary fibrosis is a progressive interstitial lung disease, which ultimately leads to respiratory failure and death. The median survival is 2-3 years and thus comparable to the survival of a malignant disease. Today, there is no cure available. Improvement of quality of life (QoL) is thus a major goal in IPF patients. Cough is a common distressing and debilitating symptom in IPF. Increased cough in IPF patients may be linked to functional upregulation of lung sensory neurones. In addition, cough independently predicts disease progression in IPF patients. Symptomatic treatment options for cough in IPF are limited. Dysregulation of the immune system has been suggested to cause IPF associated cough and treatment trials with immunomodulating agents have been promising. Unfortunately the recently studied medication thalidomide is famous for its side effects and might be apprehensively received by some patients.

Immunomodulatory effects of macrolide treatment in chronic inflammatory diseases as well as reduced cough reflex in animal studies suggest a possible reduction in cough in IPF patients. In addition, in animal in vivo models azithromycin also showed anti-fibrotic properties.

The investigators hypothesize that immunomodulatory treatment of IPF patients with AZT reduces cough frequency and might improve lung function.

Objective

The purpose of this protocol is to determine the effect of azithromycin (AZT) on subjective and objective cough, QoL and lung function, its effects on biomarkers as well as its safety in patients with idiopathic pulmonary fibrosis.Specific Objectives

1. To determine the efficiency after 12 weeks of treatment on subjective and objective cough reduction and increase of QoL
2. To monitor safety by recording severe adverse events, including mortality, organ-specific toxicities and exacerbations requiring hospitalization
3. To test efficiency at 12 weeks with overall response measured by changes in FEV1, FVC, TLC, DLCO, oxygen desaturation on exertion and 6-min walking distance
4. To determine efficiency in clinical course
5. To monitor overall adverse events
6. To determine the influence on cytokines and biomarkers in IPF
7. To determine the impact on oro-pharyngeal flora and antibiotical resistance

Methods

Single center, prospective, randomized, double blind, 2 treatments, 2 period crossover study with two 12-week treatment periods separated by a 4-week drug-free washout period and a 4 week follow-up period performed at the University Hospital Berne. All patients will be treated with both AZT and placebo. Individual changes in clinical symptoms with focus on cough frequency, life quality, lung function and adverse events will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Idiopathic pulmonary fibrosis; new diagnosis, or known. Diagnosis according to the current guidelines from ATS/ERS for IPF diagnosis, other differential diagnoses ruled out.
* Clinical symptoms of cough
* Written informed consent for study participation

Exclusion Criteria

* Previous history of an adverse reaction or allergy on azithromycin or other macrolide or ketolide antibiotics or any other ingredient (e.g. lactose)
* Evidence of respiratory infection or systemic infection one month before randomisation
* Known rhythmogenic heart disease
* Pregnancy or lactation
* History of non-compliance to medical treatment
* Current alcohol or drug abuse
* Active hepatitis, history of hepatitis, other significant liver disease
* Serum bilirubin > 50 μmol/L
* Transaminases or alkaline phosphatase elevated > 3x upper limit of normal at baseline
* Severe renal insufficiency with GFR <10ml/min
* Concomitant treatment with ergotamines
* Concomitant treatment with ciclosporin
* Concomitant treatment with ributin
* Concomitant treatment with digoxin
* Change of medication until 4 weeks before randomisation
* Pirfenidone <3 Mo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Number of patients with a subjective response to treatment | 3 months
  Subjective response is defined as a 1.3 unit reduction of cough as measured with the Leicester Cough Score from treatment start to 12 weeks of treatment.

SECONDARY OUTCOMES:
Number of patients with an objective response to treatment | 3 months
  Objective response is defined as the Overall response in the measured cough frequency by respiratory Polygraph (Resmed, Nox T3®).
Number of patients with a change in lung function | 3 months
  Measured by FEV1, FVC, TLC, & DLCO
Number of patients with a change in oxygen saturation | 3 months
  Measured by oxygen desaturation on exertion
Number of patients with a change in quality of life | 3 months
  Measured by quality of life questionnaires
Number of patients with changes in oropharyngeal flora | 3 months
Number of patients with a change in 6 min walking distance | 3 months
  Measured by oxygen desaturation on 6-min walking distance

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Funke, MD, Principal Investigator — University Hospital for Pulmonology, Berne
Locations (4):
- Switzerland (4):
  - Universitätsspital Basel, Basel
  - University Hospital for Pulmonology, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich

REFERENCES:
- [Derived] Guler SA, Clarenbach C, Brutsche M, Hostettler K, Brill AK, Schertel A, Geiser TK, Funke-Chambour M. Azithromycin for the Treatment of Chronic Cough in Idiopathic Pulmonary Fibrosis: A Randomized Controlled Crossover Trial. Ann Am Thorac Soc. 2021 Dec;18(12):2018-2026. doi: 10.1513/AnnalsATS.202103-266OC. PMID 34015241
- [Derived] Rindlisbacher B, Schmid C, Geiser T, Bovet C, Funke-Chambour M. Serum metabolic profiling identified a distinct metabolic signature in patients with idiopathic pulmonary fibrosis - a potential biomarker role for LysoPC. Respir Res. 2018 Jan 10;19(1):7. doi: 10.1186/s12931-018-0714-2. PMID 29321022
- [Derived] Rindlisbacher B, Strebel C, Guler S, Kollar A, Geiser T, Martin Fiedler G, Benedikt Leichtle A, Bovet C, Funke-Chambour M. Exhaled breath condensate as a potential biomarker tool for idiopathic pulmonary fibrosis-a pilot study. J Breath Res. 2017 Nov 29;12(1):016003. doi: 10.1088/1752-7163/aa840a. PMID 28775244